CLINICAL TRIAL: NCT03833154
Title: A Phase III, Randomized, Placebo-controlled, Double-blind, Multi-center, International Study of Durvalumab With Stereotactic Body Radiation Therapy (SBRT) for the Treatment of Patients With Unresected Stage I/II, Lymph-node Negative Non-small Cell Lung Cancer (PACIFIC-4/RTOG-3515) Osimertinib Following SBRT, a Single Arm Cohort for Patients With Unresected Stage I/II, Lymph Node Negative NSCLC Harboring a Sensitizing EGFR Mutation
Brief Title: Durvalumab With Stereotactic Body Radiation Therapy (SBRT) vs Placebo With SBRT in Early Stage Unresected Non-small Cell Lung Cancer (NSCLC) Patients/ Osimertinib Following SBRT in Patients With Early Stage Unresected NSCLC Harboring an EGFR Mutation
Acronym: PACIFIC-4
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9103C00001; 2018-002572-41 (EudraCT Number)
Record Dates: First submitted 2019-01-25; First posted 2019-02-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC; Early-Stage NSCLC; Lung cancer; Double- Blind; PD-L1; MEDI4736; Durvalumab; Osimertinib; PFS; OS; Unresected lung cancer; Medically Inoperable; Operable with Patient refusal; SBRT; SABR; EGFR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — durvalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double- Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SoC SBRT + Durvalumab Therapy (Main Cohort) (Experimental): SBRT
  Durvalumab (PD-L1 monoclonal antibody) 1500 mg every 4 weeks [q4w] intravenously [iv] for up to 26 cycles or until progression or other discontinuation criteria are met.
  Interventions: Drug: Durvalumab
- SoC SBRT + Placebo Therapy (Main Cohort) (Placebo Comparator): SBRT
  Placebo (matching placebo for infusion) every 4 weeks iv for up to 26 cycles or until progression or other discontinuation criteria are met.
  Interventions: Other: Placebo
- SoC SBRT + Osimertinib Therapy (Osimertinib cohort, single-arm, open-label separate cohort) (Experimental): SBRT
  Osimertinib 80mg every day [qd] for oral administration up to 36 months or until progression. Osimertinib treatment should start within 7 to 14 days after completion of SBRT
  Interventions: Drug: (Osimertinib cohort, single-arm, open-label separate cohort)

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500 mg every 4 weeks [q4w] intravenously [iv] for up to 26 cycles or until progression or other discontinuation criteria are met.
  Other Names: MEDI4736
  Arms: SoC SBRT + Durvalumab Therapy (Main Cohort)
Other: Placebo — Matching placebo for infusion every 4 weeks iv for up to 26 cycles or until progression or other discontinuation criteria are met.
  Arms: SoC SBRT + Placebo Therapy (Main Cohort)
Drug: (Osimertinib cohort, single-arm, open-label separate cohort) — Osimertinib 80 mg every day [qd] orally for up to 36 months or until progression or other discontinuation criteria are met. Osimertinib treatment should start from 7 to 14 days after completion of SBRT
  Arms: SoC SBRT + Osimertinib Therapy (Osimertinib cohort, single-arm, open-label separate cohort)

SUMMARY:
This is a Phase III, randomized, placebo-controlled, double-blind, multi-center study assessing the efficacy and safety of durvalumab with SoC SBRT versus placebo with SoC SBRT in patients with unresected clinical Stage I/II lymph node-negative (T1 to T3N0M0) NSCLC.

An additional cohort will assess Osimertinib following SBRT in patients with early stage unresected T1 to T3N0M0 NSCLC harbouring an EGFR mutation.

DETAILED DESCRIPTION:
Patients with Stage I/II lymph node negative NSCLC and confirmed to meet all eligibility criteria will be randomized 1:1 to receive either Durvalumab + SoC SBRT or placebo + SoC SBRT.

The primary objective of main cohort is to assess the efficacy of Durvalumab with SoC SBRT compared to placebo with SoC SBRT in terms of PFS. Key secondary is to assess the efficacy of Durvalumab with SoC SBRT compared to placebo with SoC SBRT in terms of Overall Survival (OS).

In addition, a study cohort with a sufficient number of patients harboring an EGFR-TKI sensitizing mutation, will receive Osimertinib treatment after completion of SoC SBRT as definitive treatment of Stage I/II lymph node-negative NSCLC. The primary objective of Osimertinib cohort is to assess efficacy of Osimertinib following SoC SBRT in terms of 4-year PFS. Key secondary objectives include safety, OS and efficacy of Osimertininb treatment with SBRT.

ELIGIBILITY:
Main Cohort Key Inclusion Criteria:

1. Age ≥18 years
2. Planned SoC SBRT as definitive treatment
3. World Health Organization (WHO)/ECOG PS of 0, 1 or 2
4. Life expectancy of at least 12 weeks
5. Body weight >30 kg
6. Submission of tumor tissue sample if available
7. Adequate organ and marrow function required
8. Patients with central or peripheral lesions are eligible
9. Staging studies must be done during screening (PET-CT within 10 weeks)
10. Patients with a history of metachronous NSCLC and synchronous lesions are eligible with some exceptions

Main Cohort Key Exclusion Criteria:

1. Mixed small cell and non-small cell cancer
2. History of allogeneic organ transplantation
3. History of another primary malignancy with exceptions
4. History of active primary immunodeficiency
5. Epidermal growth factor receptor local testing is strongly recommended prior to enrollment. Patients with a tumor harboring an EGFRm per local testing will be excluded from the main cohort
6. Prior exposure to immune-mediated therapy with exceptions

Osimertinib Cohort Key Inclusion Criteria

1. Age ≥18 years
2. Planned SoC SBRT as definitive treatment
3. WHO/ECOG PS of 0, 1, or 2
4. Patients with central or peripheral lesions are eligible
5. Patients with a history of metachronous NSCLC and synchronous lesions are eligible with some exceptions
6. Staging studies must be done during screening (PET-CT within 10 weeks)
7. Submission of tumor tissue sample if available
8. Confirmation by local laboratory that the tumor harbors one of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R)
9. Adequate bone marrow reserve or organ function required
10. Female patients should be using highly effective contraceptive measures
11. Male patients should be asked to use barrier contraceptives (ie, condoms) during sex with all partners during the trial and avoid procreation

Osimertinib Cohort Key Exclusion Criteria

1. Mixed small cell and non-small cell cancer
2. Patients with known or increased risk factor for QTc prolongation
3. Treatment with any of the following:

   * Preoperative or adjuvant platinum-based or other chemotherapy for the disease under investigation
   * Prior treatment with neoadjuvant or adjuvant EGFR TKI
   * Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inducers of CYP3A4
4. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of osimertinib
5. Any of the following cardiac criteria

   * Mean resting corrected QT interval >470 msec, obtained from 3 ECGs
   * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG.
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, or unexplained -sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval
   * Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) assessed by Blinded Independent Central Review (BICR) according to RECIST 1.1 in subpopulation of patients with Stage I/II NSCLC | from randomization up to 6 years
  Main Cohort
4-year Progression-Free Survival (4y-PFS) by ICR according to RECIST 1.1 criteria | from treatment start up to 5 years
  Osimertinib Cohort

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) assessed by BICR per RECIST 1.1 in all randomised patients with Stage I/II NSCLC | from randomization up to 6 years
  Main Cohort
Overall Survival (OS) | from randomization up to 7 years
  Main Cohort
Concentration of durvalumab in serum such as peak concentration and trough | 12 weeks after last dose
  Main Cohort
Detection of ADA neutralising antibodies titers | up to 6 months after last dose
  Main Cohort
Health-related quality of life in patients treated with durvalumab with SoC SBRT compared to placebo with SoC SBRT using the EORTC QLQ-C30 | from randomization up to 7 years
  Main Cohort
Proportion of patients alive and progression free at 24 months from randomisation (PFS24) assessed by BICR according to RECIST 1.1 | at 24 months following randomization
  Main Cohort
Time to progression (TTP) assessed by BICR according to RECIST 1.1 | from randomization up to 6 years
  Main Cohort
Time to death or distant metastasis (TTDM) assessed by BICR according to RECIST 1.1 | from randomization up to 6 years
  Main Cohort
Time from randomisation to second progression (PFS2) as defined by local standard clinical practice | from randomization up to 7 years
  Main Cohort
Assessment of AEs by CTCAE v 5.0 as measures of the safety and tolerability of Durvalumab with SoC SBRT compared to placebo with SoC SBRT | up to 3 months after last dose
  Main Cohort
Assessment of AEs by CTCAE v 5.0 as measures of the safety, tolerability and compliance of osimertinib with SoC SBRT therapy | Up to 35 days after last dose
  Osimertinib Cohort
WHO performance status | from treatment start up to 5 years
  Osimertinib Cohort
ECG QT interval | Up to 156 weeks of treatment or treatment discontinuation
  Osimertinib Cohort
Overall Survival | from treatment start up to 5 years
  Osimertinib Cohort
Time To Progression (TTP) | from treatment start up to 5 years
  Osimertinib Cohort
Time to CNS progression | from treatment start up to 5 years
  Osimertinib Cohort
PFS2 | from treatment start up to 5 years
  Osimertinib Cohort
Site(s) of disease progression | from treatment start up to 5 years
  Osimertinib Cohort
PFS by ICR using RECIST 1.1 | from treatment start up to 5 years
  Osimertinib Cohort

OTHER OUTCOMES:
Lung cancer mortality | from treatment start up to 5 years
  Osimertinib Cohort
Lung Cancer Mortality | from randomization Up to 5 years
  Main Cohort

CONTACTS AND LOCATIONS:
Locations (187):
- United States (74):
  - Research Site, Tuscaloosa, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Duarte, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Bay Pines, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Orlando, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Decatur, Illinois
  - Research Site, Elmhurst, Illinois
  - Research Site, Naperville, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Cedar Rapids, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, Elizabethtown, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Metairie, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, South Portland, Maine
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Rosedale, Maryland
  - Research Site, Silver Spring, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Lebanon, New Hampshire
  - Research Site, Camden, New Jersey
  - Research Site, Paramus, New Jersey
  - Research Site, Albany, New York
  - Research Site, East Syracuse, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Stony Brook, New York
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Grand Forks, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Watertown, South Dakota
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Sherman, Texas
  - Research Site, Burlington, Vermont
  - Research Site, Richmond, Virginia
  - Research Site, Bellingham, Washington
  - Research Site, Seattle, Washington
  - Research Site, Spokane Valley, Washington
  - Research Site, Milwaukee, Wisconsin
- Research Site, Clayton, Australia
- Belgium (5):
  - Research Site, Aalst
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
- Brazil (6):
  - Research Site, Barretos
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
  - Research Site, Volta Redonda
- Canada (4):
  - Research Site, Edmonton, Alberta
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (15):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Suzhou
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Zhengzhou
- France (7):
  - Research Site, Bron
  - Research Site, Dijon
  - Research Site, Lyon
  - Research Site, Nantes
  - Research Site, Pierre-Bénite
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (8):
  - Research Site, Dresden
  - Research Site, Göttingen
  - Research Site, Halle
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Homburg
  - Research Site, Regensburg
  - Research Site, Trier
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Israel (6):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (8):
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Orbassano
  - Research Site, Padua
  - Research Site, Pavia
  - Research Site, Roma
  - Research Site, Rozzano
- Japan (14):
  - Research Site, Akashi-shi
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hirosaki-shi
  - Research Site, Hiroshima
  - Research Site, Kobe
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Sunto-gun
  - Research Site, Toyoake-shi
  - Research Site, Yokohama
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Utrecht
- Poland (6):
  - Research Site, Bydgoszcz
  - Research Site, Elblag
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Lodz
  - Research Site, Warsaw
- Research Site, Hato Rey, Puerto Rico
- Russia (5):
  - Research Site, Kazan, Tatarstan
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Ufa
  - Research Site, Yekaterinburg
- South Korea (4):
  - Research Site, Cheongju-si
  - Research Site, Goyang-si
  - Research Site, Gyeonggi-do
  - Research Site, Seoul
- Spain (10):
  - Research Site, Badajoz
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, San Sebastián
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Zaragoza
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kocaeli
- United Kingdom (4):
  - Research Site, Birmingham
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Lung Cancer Study Locator details (for US) — https://www.lungcancerstudylocator.com/trial/listing/193775